CLINICAL TRIAL: NCT03696693
Title: Impact of Chronic Rhinosinusitis on the Laryngeal Mucosa and Voice Quality in Children Aged From 6- to 18- Years Old
Brief Title: Effect of Chronic Rhinosinusitis on Voice of Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Sabri Abdelraheem, principal investigator, Assiut University
Other Study IDs: rhinosinusitis in children
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Voice Disorders in Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with chronic rhinosinusitis: Children aged 6-18 years presented with symptoms of chronic rhinosinusitis will be recruited from the otorhinolaryngology out-patient clinic and department at Assiut University Hospital from October, 2018 to October, 2019.
  Interventions: Device: acoustic vocal analysis
- children without chronic rhinosinusitis: Children have the same age and number in the study group which are presented with vocal symptoms and have not chronic rhinosinusitis will be recruited for the same duration.
  Interventions: Device: acoustic vocal analysis

INTERVENTIONS:
Device: acoustic vocal analysis — Computerized Speech Laboratory (model 4300; Kay Elemetrics Corporation)
  Other Names: Video rhino- laryngoscope (3.7 mm; 8403 ZXK)

SUMMARY:
Evaluation of the effect of chronic rhinosinusitis on the laryngeal mucosa and voice quality in children. This is important to know factors affecting voice disorders

DETAILED DESCRIPTION:
The voice is that the carrier wave of verbal communication. It's created within the voice box l by vibrations of the mucous membrane of the vocal folds leading to the assembly of the first laryngeal sound. It depends on the larynx that's the voice generator, the oral fissure beside the tongue and teeth that articulate the voice, and therefore the nose with the paranasal sinuses that participate in the resonance.

Any disruption of the performance of voice is termed dysphonia. Dysphonia is outlined as perceptual audible deviation of a patient's habitual voice as self-judged or judged by his or her listeners .

"Hoarseness" or "dysphonia" are terms usually used to describe a change within the quality of the voice in which the voice are often raspy, breathy, strained, fatigued, rough, tremulous, or asthenic. There is also a change in pitch, loudness or voice breaks. The prevalence of hoarseness in children ranges from 6 to 23 percent . Boys were statistically more probably to have dysphonia (7.5%) over girls (4.6%) . the etiology of childhood dysphonia is multifactorial and factors that in previous studies have been connected to dysphonia are health- related factors , personality triats, and environmental factors . Health related factors such as recurrent inflammation of respiratory airway, Allergy and chronic cough. Personality triats such as hyperactivity and impulsiveness, besides previous history of excessive crying, Environmental factors such as pollution by noise, dryness, cold air or dust and fumes.the most common laryngeal diagnosis for children with hoarseness in a treatment - seeking population was vocal fold nodules, followed by vocal cysts, and acute laryngitis. They attribute this to vocal overuse or misuse.

Chronic rhinosinusitis is a frequently noticable condition in otorhinolaryngology clinic. 5 % to 13% of childhood viral upper airway infections may lead to acute rhinosinusitis, with a proportion of these to progress to a chronic rhinosinusitis. Chronic rhinosinusitis is defined as a minimum of ninty continuous days of two or additional symptoms of infected rhinorrhea, nasal blockage, headache, or cough and either endoscopic signs of nasal mucosal swelling and oedema, mucopurulent nasal discharge, or nasal polyposis may be associated with CT scan findings showing mucosal changes within the ostiomeatal complex and/or sinuses in a pediatric patient. The post nasal discharge is usually thick mucopurulent that goes onto the oropharyngeal and the laryngeal tissue resulting in frequent throat clearing, and cough which cause mechanical trauma and hoarse voice quality. Previous studies revealed that the voice in individuals presented with chronic sinusitis had lower values in fundamental frequency compared with those that have not sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 6 to 18 years.
* gender: both sexes will be included.
* patients with chronic rhinosinusitis according to (European Position Paper on Rhinosinusitis and Nasal Polyps 2012).

Exclusion Criteria:

* Age below 6 or above 18 years.
* Children receiving treatment for rhinosinusitis.
* Previous surgical intervention (laryngeal microsurgery or tracheal intubation).
* Congenital anomalies.
* Mental retardation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 6-18 years presented with symptoms of chronic rhinosinusitis will be recruited from the otorhinolaryngology out-patient clinic and department at Assiut University Hospital from October, 2018 to October, 2019.comparing them with children with no symptoms of chronic rhinosinusitis and complaining of vocal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
impact of chronic rhinosinusitis on the laryngeal mucosa and voice quality in children | 20 mimutes
  to evaluate effect of rhinosinusitis on acoustic voice parameters by using acoustic voice analysis (model 4300; Kay Elemetrics Corporation) and assessment changes in the laryngeal mucosa using either video rhino- laryngoscope (3.7 mm; 8403 ZXK) orRigid laryngoscope (70 degrees, 8700 CKA).

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Sabri Abd-El Raheem, PhD, Principal Investigator — Assiut University

REFERENCES:
- [Result] Develioglu ON, Paltura C, Koleli H, Kulekci M. The effect of medical treatment on voice quality in allergic rhinitis. Indian J Otolaryngol Head Neck Surg. 2013 Aug;65(Suppl 2):426-30. doi: 10.1007/s12070-013-0639-5. Epub 2013 Mar 14. PMID 24427691
- [Result] Dlova NC, Fabbrocini G, Lauro C, Spano M, Tosti A, Hift RH. Quality of life in South African Black women with alopecia: a pilot study. Int J Dermatol. 2016 Aug;55(8):875-81. doi: 10.1111/ijd.13042. Epub 2015 Nov 6. PMID 26547604
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Result] Cecil M, Tindall L, Haydon R. The relationship between dysphonia and sinusitis: a pilot study. J Voice. 2001 Jun;15(2):270-7. doi: 10.1016/S0892-1997(01)00027-3. PMID 11411480